CLINICAL TRIAL: NCT07218939
Title: Universal Biospecimen Collection Protocol for Extra Material From Clinical Pulmonary Procedures
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-1394; NCI-2025-07702 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-10-17; First posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Pulmonary

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to develop a biospecimen collection protocol for unused biospecimens from pulmonary procedures in order to facilitate research across many different areas of pulmonary medicine and mitigate the pulmonary morbidity experienced by patients with cancer.

DETAILED DESCRIPTION:
Primary objectives:

To assemble a tissue/blood bank biorepository for laboratory translational research by collecting extra samples of bronchoalveolar lavage, pleural fluid, blood or other residual tissue obtained during normally scheduled clinical procedures for the evaluation of pulmonary toxicity

To collect basic data on patient data and suspected pulmonary toxicity to cross-reference eligible biospecimens

ELIGIBILITY:
Inclusion Criteria:

All patients over the age of 18, who are seen in the Cardiopulmonary Center and are undergoing pulmonary procedures

Exclusion Criteria:

Pregnant women and prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients scheduled for pulmonary procedures in the Cardiopulmonary Center are eligible to be approached for consent and enrollment into this observational biospecimen collection protocol.
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2032-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Sheshadri, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org